CLINICAL TRIAL: NCT02844296
Title: Efficacy of a Short-bout Handgrip Exercise Intervention for Smoking Cessation: a Pilot Randomized Controlled Trial
Brief Title: Short-bout Handgrip Exercise for Smoking Cessation
Acronym: SHESC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Tung Wah Group of Hospitals (Other)
Responsible Party: Principal Investigator, Professor Lam Tai-Hing, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TWRCT2016
Record Dates: First submitted 2016-07-11; First posted 2016-07-26 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Smoking Cessation
Keywords: short-bout exercise; craving; handgrip; smoking cessation; RCT
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- exercise group (Experimental): A free handgrip (strength 15 kg) will be given to the subject and some short-bout exercise will be introduced to the subjects for reliving the cravings for smoking through a short video. After the video, the counselor will install a smartphone application which is about exercise in the subject's mobile phone to set up exercise reminder schedule for 4 weeks. 20-30 reminders on exercise and quitting tips via the App for 4 weeks. Subjects will be requested o record a daily diary on smoking.
  A leaflet with exercise instruction and motivation messages based on the Health Action Process Approach (HAPA) will be given to the participant. 2-month, 6 -month and 12-month telephone interview will be conducted. Biochemical validation will be conducted at 6-month follow up. And hand grip strength will be measured the next time when the participant comes back to CISI.
  Interventions: Behavioral: Video about exercise; Behavioral: App about exercise; Behavioral: Leaflet about exercise
- diet group (Experimental): Subjects will view a short video on healthy diet only. After the video, the counselor will also install another smartphone application which is about healthy diet in the subject's mobile phone to set up healthy die reminder schedule for 4 weeks.
  A leaflet on healthy diet will be given to the subjects, and 20-30 reminders on healthy diet and quitting tips via the App for 4 weeks.2-,6- and 12-month telephone interview will be conducted. Biochemical validation will be conducted at 6-month follow up. And hand grip strength will be measured the next time when the participant comes back to CISI.
  Interventions: Behavioral: Video about diet; Behavioral: App about diet; Behavioral: Leaflet about diet

INTERVENTIONS:
Behavioral: Video about exercise — Video about short-bout exercise will be played for the participants.
  Arms: exercise group
Behavioral: App about exercise — A smartphone App about exercise will be installed in participants' mobile phone.
  Arms: exercise group
Behavioral: Leaflet about exercise — A leaflet about exercise will be provided for the participants.
  Arms: exercise group
Behavioral: Video about diet — Video about healthy diet will be played for the participants.
  Arms: diet group
Behavioral: App about diet — A smartphone App about healthy diet will be installed in participants' mobile phone.
  Arms: diet group
Behavioral: Leaflet about diet — A leaflet about healthy diet will be provided for the participants.
  Arms: diet group

SUMMARY:
Smoking is highly addictive and quitting is difficult. Relapse is common because of withdrawal symptoms such as craving, headache, mood change and irritation. In addition to pharmacotherapy, exercise can acutely reduce craving, withdrawal symptoms and negative affect in regular smokers. Exercise effectively reduces negative affect and attentional bias towards smoking, and hence might relieve craving.Instead of long duration (30+ minutes) exercise, short-bout exercise is more easily adhered to in daily living and achieves similar health gain as long-bout exercise.Handgrip, which enhances training of hand-griping strength, is a common short-bout exercise tool used for lowering blood and arterial pressure.Therefore, this exercise tool might also raise smokers' interest to initiate this simple and effective exercise for quit attempt.

This RCT study was proposed by using short-bout exercise (intervention) and healthy diet (control ) for smoking cessation, targeting adult clients who enrolled in smoking cessation service of ICSC, smoke 10 cigarettes or more a day when they initially receive the treatment from ICSC, can access to Internet by using smart phone and interested in participating in an exercise/diet program for smoking cessation. All the participants will be randomized the subjects to one of the RCT groups by using sequentially numbered, opaque sealed envelope method. Participants from both groups will be helped to install a phone application (App) in their smartphone which can send reminders of doing exercise or healthy diet. Also, the participants will enter their smoking and craving data by the App by answering the automatic pooped daily questionnaire. Telephone follow-up will be conducted at 2,6 and 12 months.

DETAILED DESCRIPTION:
1. Scientific / historical background

   Smoking is highly addictive and quitting is difficult. Relapse is common because of withdrawal symptoms such as craving, headache, mood change and irritation. In addition to pharmacotherapy, exercise can acutely reduce craving, withdrawal symptoms and negative affect in regular smokers. Exercise effectively reduces negative affect and attentional bias towards smoking, and hence might relieve craving. A recent systematic review of the RCTs using exercise for smoking cessation suggested that more trials with larger sample size, equal contact control conditions and measures of exercise adherence are needed to confirm its effectiveness .

   Despite the effectiveness of various exercise interventions on smoking cessation, most previous RCTs required the participants to attend multiple guided exercise sessions for at least once per week consecutively for 6 to 12 weeks. Participants willing to join these sessions would have a very high motivation to quit, which might over-estimate the effect size and limit its applicability. These exercise sessions showed high compliance and effectiveness, but could only recruit very few participants who showed strong motivation to quit and had much time to attend. These interventions are unlikely to be directly applicable to the smokers in Hong Kong, who mostly prefer "self-determination" than using intensive smoking cessation services as the method of quit attempt .

   Instead of long duration (30+ minutes) exercise, short-bout exercise is more easily adhered to in daily living and achieves similar health gain as long-bout exercise . Some laboratory studies showed that short-bout (5-10 minutes) isometric exercises (e.g. jaw clenching or fist clenching) or moderate intensity exercise (e.g. stationary cycling) is effective to reduce craving and withdrawal symptoms. No published randomized controlled trials (RCT) on short-bout exercise for smoking cessation or relapse prevention from PubMed and Cochrane Library was found by the investigators.

   Handgrip, which enhances training of hand-griping strength, is a common short-bout exercise tool used for lowering blood and arterial pressure . The advantages of handgrip exercise (HGE) are: (1) The equipment is simple to use and inexpensive; (2) It can be performed anytime anywhere; (3) No intensive training is needed; (4) Effects of HGE is immediate if any on relieving craving; and (5) Adherence to HGE shall be high as it is simple to use. Grip strength has been adopted as a fitness test for recruitment into the Hong Kong Police Force, and is shown as a good predictor of cardiovascular fitness and survival. Therefore, this exercise tool might also raise smokers' interest to initiate this simple and effective exercise for quit attempt.

   Recently the research team has conducted a pilot study of delivering a short-bout exercise (about 10 minutes) intervention session using a handgrip for the clients (n=31) in the Integrated Centre on Smoking Cessation of Tung Wah Group of Hospitals and evaluating the perceived effectiveness of this exercise. In the 31 clients, 18 (59.1%) had smoking urges in the past 24 hours. Examples of the exercise were isometric griping of the handgrip as long as possible and rapid grip-and-release movements. While only 2 clients agreed that these exercises can increase abstinence before our guided exercise session, 12 post-session clients (38.7%) agreed it does. The participants perceived that the exercises are beneficial for smoking cessation, because these exercises can be conveniently performed for urge alleviation and distraction. On the other hand, the results suggested several improvements in the delivery of intervention such as increase in the exercise counselling for users with low perceived efficacy and use of handgrips with higher strength value. Applicability can be increased by incorporating other short-bout exercises, such as hand pushing and pulling, when handgrip is not available for usage. Frequency of use and increase in grip strength will be documented as indicators of exercise compliance, and additional benefits which may increase smokers' motivation.

   Short-bout exercise is a simple and low-cost behavior which only needs brief training by non-healthcare professionals and takes very little time to practice. The effect size may be small to moderate, but it has large impact as it can be disseminated easily to a large number of smokers. A short-bout exercise intervention was proposed, with handgrip mainly plus those without, to (1) reduce craving during the first month of cessation treatment and (2) increase abstinence assessed at 6-month. The main barrier of adopting such a small and easy behavior is inertia and forgetfulness. To increase the exercise adherence, Anti-inertia Reminder (AIR) model was developed and several strategies to assist the participants to overcome the inertia and forgetfulness.
2. Study design

The study consists of 3 phrases: (1a) Development of an educational video for the exercise intervention; (1b) Development of a smartphone application ("App") for reminders and electronic daily dairy; (2) Briefing session of ICSC counselors to introduce the brief short-bout exercise intervention and RCT to the clients; and (3) A randomized controlled trial to test the efficacy of delivering a brief short-bout exercise intervention for smoking cessation.

2.1 Phase 1a - Development of an educational video for the exercise intervention

2.1.1 Objective

A short video will be produced (about 5 minutes) as a part of the exercise intervention for the intervention group. It will be played in a tablet after the subjects in the intervention group have given consent to participate at recruitment. The video will also be available in the smartphone application so that he/she can watch it anytime.

2.1.2 Content

The video will (1) briefly deliver the knowledge of withdrawal symptoms during abstinence and benefits of short-bout exercise for smoking cessation; (2) guide the participants to practice the short-bout exercise, including those with or without the handgrip; (3) demonstrate the scenarios that the subject can do the exercise during work and leisure time. The handgrip is the main exercise, and the subjects should carry it along all day. Exercises without the handgrip will be demonstrated when the handgrip is not nearby; (4) advise to do the short-bout exercises as much as they can, or when they have craving.

2.2 Phase 1b - Development of a smartphone application

2.2.1 Objective

A smartphone application ("App") will be developed for automatically sending reminders of doing handgrip exercise (or healthy diet) and entering data and an electronic daily diary. All subjects will be asked to receive the reminders and enter data in the App for 4 weeks. Subjects' identification number (last 5 digits of telephone number) are entered when the App is installed on their mobile phones and used for the first time.

2.2.2 Reminder system

Subjects can set up a personalized and regular reminder schedule of exercises or diet in this App. These reminders will be short text messages with sound, pictures or vibration to motivate users to do the short-bout handgrip exercises or adopt a healthy diet. Subjects in the intervention (exercise) group will be asked to respond to these reminders by either selecting doing exercise at the moment or later. Once they select doing the exercise, a timer will be shown for timing the exercise duration. All responses to the reminders and exercise time will be recorded and uploaded to our server immediately as proxy measurements of exercise adherence. The application will generate a report showing how much handgrip exercise has been done each day by the subject so far. The sever for the App will detect if the subjects have responded the reminders, and, if not responded for a week, will notify the researchers to encourage them to try again. Subjects in the control (healthy diet) group, will not be repaired to respond the reminders, but he reminder time and data will be documented.

Subjects can also initiate the exercise timer to record the exercises anytime and anywhere. All these actions and time will be uploaded to the server.

2.2.3 Data entry of craving and smoking

All subjects in the intervention/control group will record he smoking/quitting data via the App. The App will "pop-up" a survey of 4 questions each day according to the participant's setting: (1) How many cravings do you have today? The 4 options are none, 1-2 times, 3-9 times, and every hour. (2) How is your craving in the past 24 hours? The 5 options are none, mild, fair, strong and very strong. (3) How many cigarettes do you smoke today? (4) Have you used NRT products or varenicline today? The exact time of the short survey can be set by the subject. All responses will be sent to our server and stored in the dataset immediately.

2.2.4 Other educational materials

The App will also contain the intervention videos and other relevant smoking cessation materials.

2.3 Phase 2 - Briefing session of ICSC counselors to recruit subjects to the RCT

2.3.1 Objectives

The briefing session aims to empower the ICSC service providers to (1) measure handgrip strength to encourage smokers to do exercise, (2) introduce the brief intervention of motivating the clients to practice short-bout exercise with and without handgrip, on top of their usual counselling.

2.3.2 Target service providers

All ICSC physicians, nurses, social workers and other healthcare professionals.

2.3.3 Briefing content

The two-hour briefing will include:

1. Simple motivation and empowerment of smokers to start and adhere to the exercise
2. Expected questions from smokers and suggested answers
3. Briefing on the operation of the randomized controlled trial

2.4 Phase 3 - Pilot randomized controlled trial (RCT)

2.4.1 Study design and objective

The single-blinded, 2-arm RCT aims to examine the efficacy of the short-bout exercise intervention on reducing craving and increasing tobacco abstinence.

2.4.2 Target subjects

All ICSC clients who have enrolled in the smoking cessation service will be screened by the counselor with the following eligibility criteria:

Inclusion criteria:

* Newly- or re-enrolled in the smoking cessation service of ICSC (which means existing clients are not eligible, unless they finished the previous treatment and re-enrolled)
* Consume 10 or more cigarettes when initially receive the service from ICSC
* Aged 18 years or above
* Able to communicate in Cantonese and read Chinese
* Have a smart mobile phone (IOS or Android System) with mobile internet access
* Show interest to participate in an exercise program/healthy diet for smoking cessation

Exclusion criteria:

* Incapable to do short-bout exercises due to physical or psychological conditions
* Pregnant

2.4.3 Recruitment procedures

In the 1st face-to-face session of the cessation treatment, after the usual the ICSC counselor will check the eligibility of each client for the participation of the RCT.

The counselor will briefly introduce the RCT of using short-bout exercise (treatment condition for intervention group) and healthy diet (treatment condition for control group) for smoking cessation, including follow-up schedule, and the incentives for the follow-up. If they are interested, they will be asked to sign the consent form for the participation. After the consent form, the counselor will invite them for measuring the grip strength with the dynamometer according to a standardized protocol and show the handgrip to them. Three measurements will be made for both hands of each participant. The maximum values obtained from each hand will be used for analysis.

Then, baseline information related to the socio-demographics, smoking and quitting history will be collected by the counselor (some information may have been collected in the standard baseline questionnaire of ICSC). The counselor will randomize the subject to one of the RCT groups by opening a sequentially numbered, opaque sealed envelopes (SNOSE method), followed by the intervention delivery. After the enrolment session, the counselor will immediately transfer the contact details of the participant and scan/send the documents (i. questionnaire; ii. Consent form; iii. Video feedback form via WhatsApp /Email) to the HKU research staff for follow-up. All baseline questionnaires and consent forms will be transferred to the HKU School of Public Health every 2 weeks.

2.4.4 Intervention

Intervention group

After completion of the baseline questionnaire, each subject in the intervention group will be given a free handgrip (strength 15 kg). Then, the counselor will play the short video for the participant. The intervention group will be introduced one handgrip exercise to reduce craving in the video:

* Rapid grip-and-release the handgrip for at least 30 times in 10-15 seconds in both hands,
* And short-bout exercises without handgrip will also be included: Hand pushing and pulling.

They will be encouraged to do these exercises when they have craving, or when the urge of smoking is expected. They will also be encouraged to increase the frequency and intensity of the exercise to increase the intensity to reduce craving as much as possible, and to increase their grip strength.

After the video, the counselor will assist the subject to install the App in mobile phone, set up the 4-week reminder schedule and electronic daily diary, and fill in the video feedback form. A leaflet with exercise instruction and motivation messages based on the Health Action Process Approach (HAPA) will be given to the participant.

Participants may not practice the exercise they have learned recently due to inertia, even they are interested. To break this inertia, the Anti-inertia Reminder (AIR) has been developed with several approaches in designing the intervention (1) aim to motivate each participant to do it quickly whenever they have craving, and do it every hour at least even without craving. (2) The participants are requested to make sure that the handgrip is always seen and accessible as a craving relieving "alarm". The subjects will be suggesting carry the handgrip all day and placing at an eye-catching place such as on the desk and on the dinner table. (3) Participants are required to use the smartphone application and activate the alarm setting in the 4 weeks after the baseline intervention. The participants could set a convenient time to finish the daily questionnaire. All the exercise reminders are designed based on the refined taxonomy of behavioral change techniques for physical activity in order to enhance and strength the future scientific reporting of the intervention.

Control group The control group will view a 6-minute video on healthy diet only. After the video, the counselor will also install another smartphone application which is about healthy diet in the subject's mobile phone o set up healthy die reminder schedule for 4 weeks. They will be given a leaflet on healthy diet, and 20-30 reminders on healthy diet and quitting tips via the App for 4 weeks.

Apart from all these interventions, all participants will receive usual cessation treatment in ICSC.

2.4.5 Outcomes

The primary outcomes are the 4-week self-reported smoking records for 4 weeks.

The secondary outcomes are the biochemically validated abstinence and self-reported abstinence in the past 7 days at 6-month follow up. Biochemical validated abstinence will be assessed with a Smokerlyzer, and exhaled carbon monoxide (CO) below 4ppm was defined as validated quitter. HK$50 will be offered to each client to cover their travel expense and time cost. Subjects who reported that they had quit smoking at 6-month follow up and had not use any type of nicotine replacement therapy will be invited to take a self-report biochemical validation which includes measurements of saliva cotinine. The measurement kits will be delivered to those subjects by mail. An incentive of HK$50 will then be offered to quitters who have reported the test results to the researcher. The subjects will be contacted via telephone at 2-,6- and 12-month to conduct assessment of the following outcomes : self-reported 7-day point prevalence abstinence, the Minnesota Nicotine Withdrawal Scale (MNWS) ,the International Physical Activity Questionnaire (IPAQ) , perceived effectiveness of handgrip in relieving craving (5-point Likert scale) and questionnaire of surgery drinks weekly intake. The 12-item Smoking Self-Efficacy Questionnaire (SEQ-12) will be added into the 12-month follow-up questionnaire only. Grip strength within the first two months after enrollment will be measured. Follow-ups will be measured by the ICSC counselors or HKU staff. Craving frequency, intensity and exercise adherence including frequency and duration will be entered to the App by the subjects. The mean number of days reporting smoking after craving in the 4 weeks after the enrolment, which will be assessed with 2 questions on a daily basis: (1) presence of craving (2) presence of smoking. At the enrolment, all participants will be introduced how to enter these information to the App on a daily basis during the first 4 weeks of their participation.

The 2-,6- and 12-month follow-up will be conducted when they visit the ICSC or through telephone, by a HKU research staff blinded to the group allocation. Incentive of HK$50 will be provided for their participation in each follow-up.

2.4.6 Research hypothesis

The intervention group will have a significantly greater decline of the craving frequency and intensity, a higher 4-week self-reported quit rate at 6-month follow-up than the control group, and less mean number of days reporting relapse.

2.4.7 Effect size estimation

As a pilot RCT to examine the effect size of the exercise intervention for smoking cessation, a total of 200 (each group 100) subjects will be targeted. Assuming the 6-month quit rate for the intervention and control group was 60% and 50% (based on previous data, odds ratio = 1.5), the power for the significant z-test will be 30%. The power will be 70% if the sample size is 600.

2.4.8 Randomization, allocation concealment and blinding

Simple individual randomization method by sequentially numbered, opaque sealed envelopes (SNOSE) will be used to ensure the counselors and the participants will be blinded from the allocation sequence before the group allocation. The primary investigator will prepare 384 identical, opaque, sealed, A5-sized envelops, with a unique 2-digit number with the centre name on the cover of each envelope as an identifier. Then he will create a random sequence list of the intervention or control group, and each group allocation will be sequentially numbered that is matched with the envelope identifier. A paper indicating the treatment condition will be inserted into each envelop, according to the random sequence list. The envelopes will be distributed to the 8 ICSC (48 envelopes in each ICSC). The ICSC counselor must open the envelopes following the sequence number on the envelope for the randomization procedure. The primary investigator and the HKU research staff will not be involved in the randomization of subjects.

Both the counselors and the subjects are not blinded from the behavioral intervention, but the outcome assessors (HKU research staff) at the 2- and 6-month follow-up are blinded from the group assignment.

2.4.9 Drop-out

Subjects can choose to drop out from the RCT during the study period, without any penalties or administrative procedures. If the subjects refuses to continue the intervention during the enrolment or the baseline intervention, the reasons of the drop-out should be documented by the counselor and reported to the HKU research staff on the same day. The envelopes of the drop-out participants will not be re-used for other participants.

2.4.10 Statistical analysis Data will be entered into SPSS for Windows (version 20) for analysis. By intention-to-treat (ITT) analysis and worst case scenario, participants who lost to follow-up or refused the follow-up will be treated as smokers. Chi-square tests will be used to compare categorical variables between subgroups. Complete case analysis will be done as a sensitivity analysis. Descriptive statistics including frequency, percentage, and mean will be used to summarize the outcomes and other variables. For the quitting outcomes assessed at the 2- and 6-month follow-up, logistic regression and linear regression will be used to examine the predictors. The Kolmogorov-Smirnov test will be used to determine the use of t test (normal distribution) or Mann-Whitney U test (non-normal distribution) for the comparison of continuous variables. General linear model repeated measures analysis (ANOVA) will be used to examine the changes of psychosocial variables and grip strength. To compare the number of days reporting relapse after craving in the first 4 weeks (assessed via the app) between the 2 groups, independent sample t-test will be used. For the daily outcomes including craving frequency, craving intensity and cigarette consumption (assessed via the app), linear mixed models which allow for multiple observations between subjects and account for clustering of data within subjects will be used. Both the main effect (group; exercise, for intervention group only) and interaction effect (group X day; exercise X day, for intervention group only) will be analyzed.

3. Consent

Participation in the study is voluntary. The ICSC staff at the clinics will explain to the potential subjects who agree to join the RCT that carried out RCT on smoking cessation. The smoking cessation counselors will explain to the subjects that they will receive telephone follow-ups at 2 months, 6 months and 12 months to enquire their smoking status. The subjects will be assured that they can withdraw from the study anytime without any prejudice, and all the information will be kept confidential and results will be reported in an aggregate format. Subjects are required to sign the written consent form.

4. Ethics

Ethics approval will be sought from the Institutional Review Board of the University of Hong Kong / Hong Kong Authority Hong Kong West Cluster.

5. Direct access to source data/documents

The App will only request the participants to enter research data, and the last four digital numbers of their telephone for identification. The raw data will be stored in an external hard-disk and locked in a cupboard with keys kept by the Principal Investigator. Only the Investigators and research assistant of the project will be permitted to access the raw data and/or study records. The data will be scanned and kept for 10 years or longer after the study is completed. Individual participants will not be directly identifiable from the dataset to be used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Newly- or re-enrolled in the smoking cessation service of ICSC within their first two times of visit (which means existing clients who did not enrolled the study in their first or second time of visiting the centre are not eligible, unless they finished the previous treatment and re-enrolled.)
* Consume 10 or more cigarettes when initially receive the service from ICSC
* Aged 18 years or above
* Able to communicate in Cantonese and read Chinese
* Have a smart mobile phone (IOS or Android System) with mobile internet access
* Show interest to participate in an exercise program for smoking cessation

Exclusion Criteria:

* Incapable to do short-bout exercises due to physical or psychological conditions
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
4-week self-reported tobacco abstinence at 6-month follow-up | 6 months
  4-week self-reported tobacco abstinence at 6-month follow-up

SECONDARY OUTCOMES:
Self-reported 7-day point prevalence abstinence | 2 and 6 months
  The subjects will be contacted via telephone at 2-,6-month to access: self-reported 7-day prevalence abstinence.
Grip strength measurement | baseline, 1 month and 6 months
  Grip strength (kg) at baseline, 1-month and 6-month follow-up
Minnesota Nicotine Withdrawal Scale | baseline, 2 and 6 months
  Validated Minnesota Nicotine Withdrawal Scale, which is a 5-pointed scale included 9 questions. Measured at 2-, 6- and 12-month follow-up
  Each point has a corresponding score, the scores will be added together as an overall score to predict the severity of the subject's withdrawal symptoms.
  The higher the score is, the severer the subject's withdrawal symptoms is.
International Physical Activity Questionnaire | baseline, 2 and 6 months
  The time and days of doing vigorous, moderate exercise and walking will be asked and recorded. All these exercise will be added together (Total MET-minutes/week at work = Walk (METs*min*days) + Mod (METs*min*days) + Vig(METs*min*days)).
  The higher the number the subject get, the more exercise the subject have had in the past 7 days.
Perceived effectiveness of using handgrip/healthy diet to relieve cravings for smoking | 2 months
  The subjects will be contacted via telephone at 2-month to access their perceived effectiveness of using handgrip/healthy diet to relieve cravings, which is a 5-pointed scale included 7 questions.
  Each point has a corresponding score, the scores will be added together as an overall score to predict the severity of the subject's perceived effectiveness of using handgrip/healthy diet to relieve cravings for smoking.
  The higher the score is, the more the subject's perceived handgrip/healthy diet is effective for relieving their smoking cravings.
The Smoking Self-Efficacy Questionnaire | 12 months
  The subjects will be contacted via telephone at 12-month to access the subject's self-efficacy of not smoking by using validated Smoking Self-Efficacy Questionnaire, 5-pointed scale included 13 questions.
  Each point has a corresponding score, the scores will be added together as an overall score to predict the subject's self-efficacy of not smoking.
  The higher the score is, the stronger the the subject's feel confident to not smoke.
Biochemical validated abstinence | 6 months
  Exhaled carbon monoxide will be measured with a smokerlyzer at 6 month. Participants with exhaled CO below 4ppm are defined as validated quitters.

CONTACTS AND LOCATIONS:
Overall Officials: Tai Hing Lam, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Integrated Centre on Smoking Cessation, Tung Wah Group of Hospitals, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abraham C, Michie S. A taxonomy of behavior change techniques used in interventions. Health Psychol. 2008 May;27(3):379-87. doi: 10.1037/0278-6133.27.3.379. PMID 18624603
- [Background] Badrov MB, Bartol CL, DiBartolomeo MA, Millar PJ, McNevin NH, McGowan CL. Effects of isometric handgrip training dose on resting blood pressure and resistance vessel endothelial function in normotensive women. Eur J Appl Physiol. 2013 Aug;113(8):2091-100. doi: 10.1007/s00421-013-2644-5. Epub 2013 Apr 16. PMID 23588257
- [Background] Inder JD, Carlson DJ, Dieberg G, McFarlane JR, Hess NC, Smart NA. Isometric exercise training for blood pressure management: a systematic review and meta-analysis to optimize benefit. Hypertens Res. 2016 Feb;39(2):88-94. doi: 10.1038/hr.2015.111. Epub 2015 Oct 15. PMID 26467494
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Cropsey KL, Trent LR, Clark CB, Stevens EN, Lahti AC, Hendricks PS. How low should you go? Determining the optimal cutoff for exhaled carbon monoxide to confirm smoking abstinence when using cotinine as reference. Nicotine Tob Res. 2014 Oct;16(10):1348-55. doi: 10.1093/ntr/ntu085. Epub 2014 Jun 2. PMID 24891552
- [Background] Doig GS, Simpson F. Randomization and allocation concealment: a practical guide for researchers. J Crit Care. 2005 Jun;20(2):187-91; discussion 191-3. doi: 10.1016/j.jcrc.2005.04.005. PMID 16139163
- [Background] Garg R, Malhotra V, Kumar A, Dhar U, Tripathi Y. Effect of isometric handgrip exercise training on resting blood pressure in normal healthy adults. J Clin Diagn Res. 2014 Sep;8(9):BC08-10. doi: 10.7860/JCDR/2014/8908.4850. Epub 2014 Sep 20. PMID 25386422
- [Background] Jakicic JM, Winters C, Lang W, Wing RR. Effects of intermittent exercise and use of home exercise equipment on adherence, weight loss, and fitness in overweight women: a randomized trial. JAMA. 1999 Oct 27;282(16):1554-60. doi: 10.1001/jama.282.16.1554. PMID 10546695
- [Background] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588
- [Background] Leong DP, Teo KK, Rangarajan S, Lopez-Jaramillo P, Avezum A Jr, Orlandini A, Seron P, Ahmed SH, Rosengren A, Kelishadi R, Rahman O, Swaminathan S, Iqbal R, Gupta R, Lear SA, Oguz A, Yusoff K, Zatonska K, Chifamba J, Igumbor E, Mohan V, Anjana RM, Gu H, Li W, Yusuf S; Prospective Urban Rural Epidemiology (PURE) Study investigators. Prognostic value of grip strength: findings from the Prospective Urban Rural Epidemiology (PURE) study. Lancet. 2015 Jul 18;386(9990):266-73. doi: 10.1016/S0140-6736(14)62000-6. Epub 2015 May 13. PMID 25982160
- [Background] Leung DY, Chan SS, Lau CP, Wong V, Lam TH. An evaluation of the psychometric properties of the Smoking Self-Efficacy Questionnaire (SEQ-12) among Chinese cardiac patients who smoke. Nicotine Tob Res. 2008 Aug;10(8):1311-8. doi: 10.1080/14622200802238928. PMID 18686178
- [Background] Michie S, Ashford S, Sniehotta FF, Dombrowski SU, Bishop A, French DP. A refined taxonomy of behaviour change techniques to help people change their physical activity and healthy eating behaviours: the CALO-RE taxonomy. Psychol Health. 2011 Nov;26(11):1479-98. doi: 10.1080/08870446.2010.540664. Epub 2011 Jun 28. PMID 21678185
- [Background] Roberts V, Maddison R, Simpson C, Bullen C, Prapavessis H. The acute effects of exercise on cigarette cravings, withdrawal symptoms, affect, and smoking behaviour: systematic review update and meta-analysis. Psychopharmacology (Berl). 2012 Jul;222(1):1-15. doi: 10.1007/s00213-012-2731-z. Epub 2012 May 15. PMID 22585034
- [Background] Taylor AH, Ussher MH, Faulkner G. The acute effects of exercise on cigarette cravings, withdrawal symptoms, affect and smoking behaviour: a systematic review. Addiction. 2007 Apr;102(4):534-43. doi: 10.1111/j.1360-0443.2006.01739.x. PMID 17286639
- [Background] Ussher M, Cropley M, Playle S, Mohidin R, West R. Effect of isometric exercise and body scanning on cigarette cravings and withdrawal symptoms. Addiction. 2009 Jul;104(7):1251-7. doi: 10.1111/j.1360-0443.2009.02605.x. PMID 19563567
- [Background] Ussher M, Nunziata P, Cropley M, West R. Effect of a short bout of exercise on tobacco withdrawal symptoms and desire to smoke. Psychopharmacology (Berl). 2001 Oct;158(1):66-72. doi: 10.1007/s002130100846. PMID 11685385
- [Background] Ussher M, West R, Doshi R, Sampuran AK. Acute effect of isometric exercise on desire to smoke and tobacco withdrawal symptoms. Hum Psychopharmacol. 2006 Jan;21(1):39-46. doi: 10.1002/hup.744. PMID 16389665
- [Background] Van Rensburg KJ, Taylor A, Hodgson T. The effects of acute exercise on attentional bias towards smoking-related stimuli during temporary abstinence from smoking. Addiction. 2009 Nov;104(11):1910-7. doi: 10.1111/j.1360-0443.2009.02692.x. PMID 19832788
- [Background] Yu X, Xiao D, Li B, Liu Y, Wang G, Chen J, Bai C, Pan J, Wan H, Li Q, Zhou X, Liao R, Li Q, Wang C, Chen R, Tang Y, Mo H, Zhao M, Du J, Li J, Kang L, Wang C. Evaluation of the Chinese versions of the Minnesota nicotine withdrawal scale and the questionnaire on smoking urges-brief. Nicotine Tob Res. 2010 Jun;12(6):630-4. doi: 10.1093/ntr/ntq063. Epub 2010 May 24. PMID 20498226
- [Derived] Cheung YT, Lam TH, Chan CHH, Ho KS, Fok WYP, Wang MP, Li WHC. Brief handgrip and isometric exercise intervention for smoking cessation: A pilot randomized trial. Addict Behav. 2020 Jan;100:106119. doi: 10.1016/j.addbeh.2019.106119. Epub 2019 Sep 4. PMID 31522134